CLINICAL TRIAL: NCT02300142
Title: Rollover Trial for Placebo Subjects Previously Enrolled Into GEN-003-002 - Randomized, Double-Blind, Factorial Study to Compare the Safety and Efficacy of Combinations of GEN-003 and Matrix-M2 in Subjects With Genital HSV-2
Brief Title: Rollover Trial for Placebo Subjects Previously Enrolled Into GEN-003-002 Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genocea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GEN-003-002a
Record Dates: First submitted 2014-11-20; First posted 2014-11-24 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Genital Herpes Simplex Type 2
Keywords: HSV; Herpes; genital infection; vaccine
MeSH Terms: conditions — Herpes Simplex | interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- GEN-003 Vaccine 30μg / Matrix-M 25μg (Experimental): GEN-003 Vaccine (30 μg of each antigen) with Matrix-M2 adjuvant (25 μg), administered as a 0.5 mL intramuscular (IM) injection.
  Interventions: Biological: GEN-003 Vaccine (30μg of each antigen); Biological: Matrix-M2 Adjuvant (25μg)
- GEN-003 Vaccine 30μg / Matrix-M2 50μg (Experimental): GEN-003 Vaccine (30 μg of each antigen) with Matrix-M2 adjuvant (50 μg), administered as a 0.5 mL intramuscular (IM) injection.
  Interventions: Biological: GEN-003 Vaccine (30μg of each antigen); Biological: Matrix-M2 Adjuvant (50μg)
- GEN-003 Vaccine 30μg / Matrix-M2 75μg (Experimental): GEN-003 Vaccine (30 μg of each antigen) with Matrix-M2 adjuvant (75 μg), administered as a 0.5 mL intramuscular (IM) injection.
  Interventions: Biological: GEN-003 Vaccine (30μg of each antigen); Biological: Matrix-M2 Adjuvant (75μg)
- GEN-003 Vaccine 60μg / Matrix-M2 25μg (Experimental): GEN-003 Vaccine (60 μg of each antigen) with Matrix-M2 adjuvant (25 μg), administered as a 0.5 mL intramuscular (IM) injection.
  Interventions: Biological: GEN-003 Vaccine (60μg of each antigen); Biological: Matrix-M2 Adjuvant (25μg)
- GEN-003 Vaccine 60μg / Matrix-M2 50μg (Experimental): GEN-003 Vaccine (60 μg of each antigen) with Matrix-M2 adjuvant (50 μg), administered as a 0.5 mL intramuscular (IM) injection.
  Interventions: Biological: GEN-003 Vaccine (60μg of each antigen); Biological: Matrix-M2 Adjuvant (50μg)
- GEN-003 Vaccine 60μg / Matrix-M2 75μg (Experimental): GEN-003 Vaccine (60 μg of each antigen) with Matrix-M2 adjuvant (75 μg), administered as a 0.5 mL intramuscular (IM) injection.
  Interventions: Biological: GEN-003 Vaccine (60μg of each antigen); Biological: Matrix-M2 Adjuvant (75μg)

INTERVENTIONS:
Biological: GEN-003 Vaccine (30μg of each antigen) — HSV-2 protein subunit vaccine consisting of 2 recombinant T cell antigens: internal fragment of the immediate early (IE) protein ICP and glycoprotein D
  Other Names: HSV Vaccine
  Arms: GEN-003 Vaccine 30μg / Matrix-M 25μg; GEN-003 Vaccine 30μg / Matrix-M2 50μg; GEN-003 Vaccine 30μg / Matrix-M2 75μg
Biological: GEN-003 Vaccine (60μg of each antigen) — HSV-2 protein subunit vaccine consisting of 2 recombinant T cell antigens: internal fragment of the immediate early (IE) protein ICP and glycoprotein D
  Other Names: HSV Vaccine
  Arms: GEN-003 Vaccine 60μg / Matrix-M2 25μg; GEN-003 Vaccine 60μg / Matrix-M2 50μg; GEN-003 Vaccine 60μg / Matrix-M2 75μg
Biological: Matrix-M2 Adjuvant (25μg) — Matrix-M2 is derived from fractionated Quillaja saponins, phosphatidylcholine, and cholesterol.
  Other Names: MM2; Adjuvant
  Arms: GEN-003 Vaccine 30μg / Matrix-M 25μg; GEN-003 Vaccine 60μg / Matrix-M2 25μg
Biological: Matrix-M2 Adjuvant (50μg) — Matrix-M2 is derived from fractionated Quillaja saponins, phosphatidylcholine, and cholesterol.
  Other Names: MM2; Adjuvant
  Arms: GEN-003 Vaccine 30μg / Matrix-M2 50μg; GEN-003 Vaccine 60μg / Matrix-M2 50μg
Biological: Matrix-M2 Adjuvant (75μg) — Matrix-M2 is derived from fractionated Quillaja saponins, phosphatidylcholine, and cholesterol.
  Other Names: MM2; Adjuvant
  Arms: GEN-003 Vaccine 30μg / Matrix-M2 75μg; GEN-003 Vaccine 60μg / Matrix-M2 75μg

SUMMARY:
This is a voluntary study to allow subjects who received placebo while on GEN-003-002 to be randomized, in a blinded manner, to 1 of 6 active combinations of GEN-003 and Matrix-M2.

Objectives:

* To compare the impact on clinical Herpes Simplex Virus type-2 (HSV-2) disease among 6 different combinations of GEN-003 antigens and Matrix-M2 adjuvant measured by:

  * Time to first clinical and/or virologic recurrence after Dose 3 (Day 43)
  * Proportion of subjects who are recurrence free at 6 and 12 months after the last dose of vaccine
  * Lesion rate (percent of days with genital lesions present) during the post-vaccination follow-up period
  * Antiviral use.
* To evaluate the safety and tolerability of GEN-003 in combination with Matrix-M2.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who received placebo in GEN-003-002 and completed the study through Day 71 per protocol, including the collection of at least 45 anogenital swabs during Days 43 to 71.
2. Enrolled into this trial within 56 days of completing Day 71 of GEN-003-002.
3. Willing and able to provide written informed consent.
4. Willing to perform and comply with all study procedures including attending clinic visits as scheduled.
5. Men and women of childbearing potential, must be willing to practice a highly effective method of contraception that may include, but is not limited to, abstinence, monogamous relationship with vasectomized partner, vasectomy, licensed hormonal methods, intrauterine device (IUD), or barrier method (e.g., condom, diaphragm) for 28 days before and 90 days after receiving Study Drug.

Exclusion Criteria:

1. On suppressive antiviral medication within 7 days prior to the first dose of Study Drug.
2. Collection of less than 45 anogenital swabs during Days 43 to 71 of the GEN-003-002 study.
3. History of any form of ocular Herpes Simplex Virus (HSV) infection, HSV-related erythema multiforme, or herpes meningitis or encephalitis.
4. Immunocompromised individuals, including those receiving immunosuppressive doses of corticosteroids (more than 20 mg of prednisone given daily or on alternative days for 2 weeks or more within 6 months prior to the first dose of Study Drug, any dose of corticosteroids within 30 days of the first dose of Study Drug, or high dose inhaled corticosteroids [> 960 μg/day of beclomethasone dipropionate or equivalent]) or other immunosuppressive agents.
5. Presence or history of autoimmune disease, regardless of current treatment.
6. Positive serologic test for Human Immunodeficiency Virus (HIV-1) or hepatitis C infection (in the absence of a negative PCR result); positive hepatitis B surface antigen (HBsAg) within 6 months prior to the first dose of Study Drug.
7. Clinically significant laboratory abnormality or a value ≥ Grade 2 within 56 days prior to the first dose of Study Drug.
8. Receipt of blood products within 90 days prior to the first dose of Study Drug.
9. Receipt of a live vaccine within 28 days prior to or a subunit vaccine within 14 days prior to the first dose of Study Drug or planned vaccination within 30 days following the last dose of Study Drug.
10. Pregnant or nursing women.
11. History of drug or alcohol abuse that, in the opinion of the Investigator, would interfere with the patient's ability to comply with the requirements of the study.
12. Other active, uncontrolled co-morbidities that, in the opinion of the Investigator, would make the subject unsuitable for the study or unable to comply with the study requirements.

NOTE: Subjects who are taking a medication to control an underlying co-morbidity may be enrolled if there have been no changes to their medication within 60 days prior to the first dose of Study Drug.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Impact on clinical HSV-2 disease based on time to recurrence and lesion rate | 53 weeks

SECONDARY OUTCOMES:
Number of patients with adverse events as a measure of safety and tolerability | 57 weeks

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - University of Alabama Vaccine Research Unit, Birmingham, Alabama
  - Medical Center for Clinical Research, San Diego, California
  - Quest Clinical Research, San Francisco, California
  - University of Illinois Department of Medicine, Chicago, Illinois
  - Indiana University Infectious Disease Research, Indianapolis, Indiana
  - The Fenway Institute, Boston, Massachusetts
  - UNC Global HIV Prevention and Treatment Clinical Trials Unit, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Westover Heights Clinic, Portland, Oregon
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Tekton Research, Austin, Texas
  - Center for Clinical Studies - Houston, Houston, Texas
  - Center for Clinical Studies, Houston, Texas
  - Center for Clinical Studies - Clear Lake/Webster, Webster, Texas
  - University of Utah, Salt Lake City, Utah
  - UW Virology Research Clinic, Seattle, Washington